CLINICAL TRIAL: NCT01030575
Title: Phase II Randomized, Double-Masked, Placebo-Controlled, Safety, Pharmacokinetic, and Dose-Ranging Study of Multiple Doses of Inositol in Premature Infants
Brief Title: Multi-dose Pharmacokinetics and Dose Ranging of Inositol in Premature Infants (INS-2)
Acronym: INS-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Eye Institute (NEI) (NIH); National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NICHD-NRN-0036-2; U10HD021364 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027871 (NIH); U10HD027880 (NIH); U10HD027904 (NIH); U10HD034216 (NIH); U10HD036790 (NIH); U10HD040492 (NIH); U10HD040689 (NIH); U10HD053089 (NIH); U10HD053109 (NIH); U10HD053119 (NIH); U10HD053124 (NIH); UL1RR024139 (NIH); UL1RR025744 (NIH); UL1RR024979 (NIH); M01RR008084 (NIH)
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Results first posted 2021-03-12 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-03

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Retinopathy of Prematurity; Bronchopulmonary Dysplasia (BPD)
Keywords: NICHD Neonatal Research Network; Pharmacokinetics; Inositol; Very Low Birth Weight (VLBW); Extremely Low Birth Weight (ELBW); Prematurity
MeSH Terms: conditions — Premature Birth; Retinopathy of Prematurity; Bronchopulmonary Dysplasia | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Inositol low volume (Experimental): 10 mg/kg/day Intravenous inositol 5%
  Interventions: Drug: Inositol lower volume
- Inositol mid-level volume (Experimental): 40 mg/kg/day Intravenous inositol 5%
  Interventions: Drug: Inositol mid-level volume
- Inositol high volume (Experimental): 80 mg/kg/day Intravenous inositol 5%
  Interventions: Drug: Inositol high volume
- Placebo (Placebo Comparator): Glucose 5% given in volumes equal to that of the comparator drug
  Interventions: Drug: Placebo low volume

INTERVENTIONS:
Drug: Inositol lower volume — 5 mg/kg/dose inositol every 12 hours, given intravenously over 20 minutes
  Other Names: Myo-inositol 5%
  Arms: Inositol low volume
Drug: Inositol mid-level volume — 20 mg/kg/dose inositol every 12 hours, given intravenously over 20 minutes
  Other Names: Myo-inositol 5%
  Arms: Inositol mid-level volume
Drug: Inositol high volume — 40 mg/kg/dose inositol every 12 hours, given intravenously over 20 minutes
  Other Names: Myo-inositol 5%
  Arms: Inositol high volume
Drug: Placebo low volume — Glucose 5% given in volumes equal to that of the comparator drug
  Other Names: Dextrose
  Arms: Placebo

SUMMARY:
This pilot study is a randomized, placebo-controlled, clinical trial to measure changes in blood and urine levels of inositol in premature infants at high risk for retinopathy of prematurity (ROP) following repeated doses of inositol. Based on previous studies, the premise is that maintaining inositol concentrations similar to those occurring naturally in utero will reduce the rates of ROP and bronchopulmonary dysplasia in premature infants. The objective is to evaluate pharmacokinetics, safety, and clinical outcomes of multiple doses of three different dose amounts of myo-inositol (provided by Abbott Laboratories) in very low birth weight premature infants. This study will enroll an estimated 96 infants at 17 NICHD Neonatal Research Network sites. Infants will be randomly assigned to receive either 10 mg/kg of 5% inositol, 40 mg/kg of 5% inositol, 80 mg/kg of 5% inositol, or 5% glucose given in the same volumes and timings as the inositol dosage to maintain masking. Enrollees will receive their assigned dose or placebo daily, starting within 72 hours of birth, and continuing until they reach 34 weeks post-menstrual age, 10 weeks chronologic age, or until the time of hospital discharge, whichever occurs first. The study drug will be administered first intravenously; as the infants progress to full feeding, the drug will be given enterally (orally or via feeding tube). Enrollees will be seen for a follow-up examination at 18-22 months corrected age. This pilot study is in preparation for a future Phase III multi-center randomized controlled trial.

DETAILED DESCRIPTION:
Retinopathy of prematurity (ROP) is an abnormal growth of the blood vessels in the eye that occurs primarily in very premature infants. Eye development occurs normally in the womb; in infants born prematurely, however, the blood vessels must finish developing outside the protective environment of the uterus. Retinopathy of prematurity (also known as retrolental fibroplasia) is a leading cause of blindness and other vision impairments (myopia, strabismus, and amblyopia) in children, both in developed and developing countries.

Inositol is a naturally-occurring sugar alcohol produced by the fetus and placenta and is present in high levels in fetal blood throughout pregnancy in humans and other animals. Serum levels fall rapidly after birth, although this fall is moderated in infants who receive breast milk or fortified formula. Two randomized trials have shown that intravenous inositol supplementation in the first week significantly reduced death, bronchopulmonary dysplasia (BPD), and retinopathy. One study of enteral supplements (given orally or via feeding tube) was less convincing, but also supported reduction of retinopathy.

This pilot study will evaluate changes in blood and urine inositol levels (half-life pharmacokinetics) of multiple doses of myo-inositol (provided by Abbott Laboratories, Abbott Nutrition Division) given to very low birth weight infants. The premise is that maintaining inositol concentrations similar to those occurring naturally in utero will reduce the rates of retinopathy and bronchopulmonary dysplasia in premature infants. Results from this study will be used to select the dose for a large multi-center trial.

In this study, 17 NICHD Neonatal Research Network sites will enroll approximately 96 infants at 12-72 hours of age. Enrolled infants will be randomly assigned to receive either 10mg/kg of 5% inositol, 40 mg/kg of 5% inositol, 80 mg/kg of 5% inositol, or 5% glucose given in the same volumes and timings as the inositol dosage to maintain masking. Inositol will be administered intravenously until babies are feeding normally, at which time the same dose and formulation will be administered enterally (orally or via feeding tube). Concentrations of inositol will be measured in blood, urine, and milk received.

Stratification: Recruitment will be stratified by gestational age into infants born at 23 0/7 to 26 6/7 weeks gestational age and infants born at 27 0/7 to 29 6/7 weeks gestational age.

ELIGIBILITY:
Inclusion Criteria:

* 23 0/7 to 26 6/7 weeks gestational age (48 infants) or
* 27 0/7 to 29 6/7 weeks gestational age (48 infants)
* 401 grams birth weight or larger
* 12-72 hours of age

Exclusion Criteria:

* Major congenital and intracranial anomalies
* Moribund or not to be provided continued support
* Seizures
* Suspected renal failure (oliguria <0.6 cc/kg/hr for >24 hours or creatinine >2.5 mg/dL)

Ages: 12 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abbot R. Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Michele C. Walsh, MD MS, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Ronald N. Goldberg, MD, Principal Investigator — Duke University; Barbara J. Stoll, MD, Principal Investigator — Emory University; Brenda B. Poindexter, MD MS, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P. Van Meurs, MD, Principal Investigator — Stanford University; Ivan D. Frantz III, MD, Principal Investigator — Tufts Medical Center; Kurt Schibler, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Edward F Bell, MD, Principal Investigator — University of Iowa; Kristi L. Watterberg, MD, Principal Investigator — University of New Mexico; Dale L. Phelps, MD, Principal Investigator — University of Rochester; Pablo J. Sanchez, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Kathleen A. Kennedy, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Roger G. Faix, MD, Principal Investigator — University of Utah; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NDASG

REFERENCES:
- [Result] Phelps DL, Ward RM, Williams RL, Nolen TL, Watterberg KL, Oh W, Goedecke M, Ehrenkranz RA, Fennell T, Poindexter BB, Cotten CM, Hallman M, Frantz ID 3rd, Faix RG, Zaterka-Baxter KM, Das A, Ball MB, Lacy CB, Walsh MC, Carlo WA, Sanchez PJ, Bell EF, Shankaran S, Carlton DP, Chess PR, Higgins RD. Safety and pharmacokinetics of multiple dose myo-inositol in preterm infants. Pediatr Res. 2016 Aug;80(2):209-17. doi: 10.1038/pr.2016.97. Epub 2016 Apr 13. PMID 27074126
- See also: NICHD Neonatal Research Network — https://neonatal.rti.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants who were 23(0/7) to 29(6/7) weeks gestational age, weighed at least 400grams, survived >12 hours, and could receive study drug by 72 hours after birth were screened and enrolled (after meeting eligibility criteria) across 14 centers of the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Neonatal Research Network (NRN)
Period: Overall Study
Arm/Group | Inositol Low Volume | Inositol Mid-level Volume | Inositol High Volume | Placebo
Started (3 infants were randomized but did not receive treatment; 2 died and 1 was determined ineligible.) | 29 | 30 | 28 | 35
Completed | 29 (1 infant randomized to the placebo arm incorrectly received the low dose. The infant was included in the low dose arm for the pharmacokinetics analyses and as randomized to the placebo arm for all other analyzes.) | 30 | 28 | 35 (1 infant randomized to the placebo arm incorrectly received the low dose. The infant was included in the low dose arm for the pharmacokinetics analyses and as randomized to the placebo arm for all other analyzes.)
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inositol Low Volume | Inositol Mid-level Volume | Inositol High Volume | Placebo | Total
Number analyzed (Participants) | 29 | 30 | 28 | 35 | 122
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Gestational Age
  weeks | 26.6 (1.8) | 26.7 (1.8) | 26.7 (1.9) | 26.5 (1.6) | 26.6 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 16 | 17 | 62
  Male | 14 | 16 | 12 | 18 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 8 | 9 | 27
  Not Hispanic or Latino | 26 | 23 | 20 | 26 | 95
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 0 | 0 | 3
  Asian | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 15 | 12 | 13 | 18 | 58
  White | 9 | 17 | 15 | 17 | 58
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Head Circumference [Mean (Standard Deviation); unit: cm] | 24.1 (2.0) | 25.1 (2.5) | 24.6 (1.9) | 23.8 (2.0) | 24.3 (2.1)
Birth Weight [Mean (Standard Deviation); unit: grams] | 897 (272) | 939 (245) | 921 (286) | 884 (224) | 909 (253)
Antenatal Steroids [Count of Participants; unit: Participants]
  Yes | 24 | 24 | 26 | 32 | 106
  No | 5 | 6 | 2 | 3 | 16
Early Onset Sepsis [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 0 | 0 | 1
  No | 29 | 29 | 28 | 35 | 121
Cesarean Delivery [Count of Participants; unit: Participants]
  Yes | 16 | 19 | 14 | 21 | 70
  No | 13 | 11 | 14 | 14 | 52
Chorioamnionitis [Count of Participants; unit: Participants]
  Yes | 4 | 4 | 3 | 5 | 16
  No | 25 | 26 | 25 | 30 | 106
APGAR 1-minute [Median (Full Range); unit: units on a scale] — APGAR score range is 1 to 10; higher scores indicate the baby is doing better immediately after birth. A: Activity/muscle tone (0-2 points): P: Pulse/heart rate (0-2 points); G: Grimace (0-2 points); A: Appearance (0-2 points); R: Respiration/breathing (0-2 points)
  units on a scale | 5 [1 to 8] | 3 [1 to 8] | 5 [1 to 8] | 3 [1 to 9] | 4 [1 to 9]
APGAR 5-minute [Median (Full Range); unit: units on a scale] — APGAR score range is 1 to 10; higher scores indicate the baby is doing better immediately after birth. A: Activity/muscle tone (0-2 points): P: Pulse/heart rate (0-2 points); G: Grimace (0-2 points); A: Appearance (0-2 points); R: Respiration/breathing (0-2 points)
  units on a scale | 8 [1 to 9] | 7 [1 to 8] | 7 [3 to 9] | 7 [1 to 9] | 7 [1 to 9]
Gestational Age (GA) STRATUM [Count of Participants; unit: Participants]
  23-26 Weeks | 15 | 16 | 14 | 19 | 64
  27-29 Weeks | 14 | 14 | 14 | 16 | 58

OUTCOME MEASURES:

1. Primary Outcome: Population Pharmacokinetics: V - Volume
Time Frame: 8-10 blood samples per infant were drawn over 10 weeks for infant safety with the full study duration represented across all infants. Samples were drawn at baseline & on days 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, 28, 35, 42, 56, and 70.
Population: All 4 arms of the study are used in the Pop-PK analysis population. 1 infant randomized to the placebo arm incorrectly received the low dose. The infant was included in the low dose arm for the pharmacokinetics analyses and as randomized to the placebo arm for all other analyzes.
Measure: Mean (Standard Error); unit: l/kg
Groups:
- PK Population: A population pharmacokinetics (Pop-PK) model was used to combine the serum inositol concentrations measured at the sparse sampling time points described under Time Frame. A 1-compartment multiple-administration intravenous infusion model with linear elimination and an added term for a steady state infusion rate of inositol from feeding and endogenous synthesis. The model is used to estimate typical (fixed effect) values of volume of distribution (V), clearance (Cl) and endogenous infusion rate (R). It is not possible to include separate estimates of the Pop-PK parameters by arm since the same values are used across all arms combined with the dosage of inositol received by an infant applied separately in the Pop-PK model.
Arm/Group | PK Population
Number analyzed (Participants) | 122
l/kg | 0.6572 (0.0707)

2. Primary Outcome: Population Pharmacokinetics: Cl - Clearance
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: (l/kg)/h
Arm/Group | PK Population
Number analyzed (Participants) | 122
(l/kg)/h | 0.0577 (0.0061)

3. Primary Outcome: Population Pharmacokinetics: R - Endogenous Infusion Rate
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: (mg/kg)/h
Arm/Group | PK Population
Number analyzed (Participants) | 122
(mg/kg)/h | 2.369 (0.3151)

4. Primary Outcome: Population Pharmacokinetics: k - Elimination Rate (Cl/V)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: liter/hour
Arm/Group | PK Population
Number analyzed (Participants) | 122
liter/hour | 0.0878 (0.0137)

5. Primary Outcome: Population Pharmacokinetics: t1/2 - Half-Life (0.693/k)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: hour
Arm/Group | PK Population
Number analyzed (Participants) | 122
hour | 7.90 (1.229)

6. Primary Outcome: Population Pharmacokinetics: E - Concentration Due to Endogenous Infusion (R/Cl)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: miligrams/liter
Arm/Group | PK Population
Number analyzed (Participants) | 122
miligrams/liter | 41.06 (1.777)

7. Primary Outcome: SD of Residual Error (mg/l)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/l
Arm/Group | PK Population
Number analyzed (Participants) | 122
mg/l | 24.77 (0.971)

8. Secondary Outcome: Number of Participants With Any Retinopathy of Prematurity (ROP)
Description: Any ROP is defined as ROP of any severity that is observed at 18-22 month corrected age
Time Frame: 18-22 month corrected age
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Inositol Low Volume | Inositol Mid-level Volume | Inositol High Volume | Placebo
Number analyzed (Participants) | 24 | 23 | 25 | 24
Participants | 11 | 11 | 14 | 12

9. Secondary Outcome: Number of Participants With Any Retinopathy of Prematurity Through 18-22 Month Corrected Age or Death
Description: Number of participants with any Retinopathy of Prematurity (ROP) through 18-22 month corrected age or death
Time Frame: 18-22 month corrected age
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Inositol Low Volume | Inositol Mid-level Volume | Inositol High Volume | Placebo
Number analyzed (Participants) | 26 | 29 | 26 | 30
Participants | 13 | 17 | 15 | 18

10. Secondary Outcome: Number of Participants With Any Ophthalmologic Diagnosis
Description: Any ophthalmologic diagnosis at 18-22 month corrected age
Time Frame: 18-22 month corrected age
Measure: Count of Participants; unit: Participants
Arm/Group | Inositol Low Volume | Inositol Mid-level Volume | Inositol High Volume | Placebo
Number analyzed (Participants) | 24 | 21 | 22 | 21
Participants | 9 | 6 | 10 | 5

11. Secondary Outcome: Number of Participants With Any Ophthalmologic Treatment
Description: Any ophthalmologic treatment at 18-22 month corrected age
Time Frame: 18-22 month corrected age
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Inositol Low Volume | Inositol Mid-level Volume | Inositol High Volume | Placebo
Number analyzed (Participants) | 24 | 21 | 22 | 21
Participants | 4 | 4 | 2 | 5

12. Secondary Outcome: Number of Participants With Any Ophthalmologic Surgical Treatment
Description: Any ophthalmologic surgical treatment at 18-22 month corrected age
Time Frame: 18-22 month corrected age
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Inositol Low Volume | Inositol Mid-level Volume | Inositol High Volume | Placebo
Number analyzed (Participants) | 24 | 21 | 22 | 21
Participants | 3 | 4 | 0 | 4

13. Secondary Outcome: Number of Participants With Any Ophthalmologic Medical Treatment
Description: Any ophthalmologic medical treatment at 18-22 month corrected age
Time Frame: 18-22 month corrected age
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Inositol Low Volume | Inositol Mid-level Volume | Inositol High Volume | Placebo
Number analyzed (Participants) | 24 | 21 | 22 | 21
Participants | 2 | 1 | 1 | 2

14. Secondary Outcome: Number of Participants With Moderate or Severe Neurodevelopmental Impairment at 18-22 Month Corrected Age
Description: A composite outcome that measures the occurrence of neurodevelopmental impairment between birth and 18-22 months corrected age.
Time Frame: 18-22 month corrected age
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Inositol Low Volume | Inositol Mid-level Volume | Inositol High Volume | Placebo
Number analyzed (Participants) | 24 | 23 | 22 | 27
Participants | 8 | 9 | 11 | 13

15. Secondary Outcome: Number of Participants With Moderate or Severe Neurodevelopmental Impairment at 18-22 Month Corrected Age or Death
Description: Moderate or Severe NDI defined as occurrence of any of the following: GMFCS level II or higher (severe is level 4 or 5), Bayley III cognitive composite score < 85 (severe is <70), Bayley III motor composite score < 85 (severe is <70), unilateral blind or bilateral blind, permanent hearing loss that does not permit child to understand directions of the examiner and communicate despite amplification with cochlear implant or hearing aid
Time Frame: 8-22 months corrected age.
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Inositol Low Volume | Inositol Mid-level Volume | Inositol High Volume | Placebo
Number analyzed (Participants) | 26 | 29 | 24 | 34
Participants | 10 | 15 | 13 | 20

16. Secondary Outcome: Number of Participants With Moderate or Severe Cerebral Palsy
Description: Cerebral palsy by severity category (absent/mild/moderate/severe).
Time Frame: 18-22 months corrected age.
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Inositol Low Volume | Inositol Mid-level Volume | Inositol High Volume | Placebo
Number analyzed (Participants) | 24 | 24 | 23 | 27
Participants | 0 | 1 | 1 | 2

17. Secondary Outcome: Number of Participants With Composite Motor Score Less Than 70
Description: This is measured as a scored of less than 70 on the Bayley Scale of Infant and Toddler Development (BSID)-III composite motor score. Higher scores indicate better performance.
Time Frame: 18-22 months corrected age
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Inositol Low Volume | Inositol Mid-level Volume | Inositol High Volume | Placebo
Number analyzed (Participants) | 24 | 22 | 22 | 25
Participants | 1 | 1 | 2 | 6

18. Secondary Outcome: Number of Participants With Composite Cognitive Score Less Than 70
Description: This is measured as a score of less than 70 on the Bayley Scale of Infant and Toddler Development (BSID)-III composite cognitive score
Time Frame: 18-22 months corrected age.
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Inositol Low Volume | Inositol Mid-level Volume | Inositol High Volume | Placebo
Number analyzed (Participants) | 24 | 23 | 22 | 26
Participants | 0 | 1 | 1 | 2

19. Secondary Outcome: Number of Participants With Severe Hearing Impairment
Description: Defined as permanent hearing loss that does not permit child to understand directions of the examiner and communicate despite amplification with cochlear implant or hearing aid.
Time Frame: 18-22 months corrected age.
Population: Intent to Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Inositol Low Volume | Inositol Mid-level Volume | Inositol High Volume | Placebo
Number analyzed (Participants) | 24 | 24 | 23 | 27
Participants | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Severe Vision Loss
Description: Vision loss as diagnosed by an ophthalmologist as legally blind, and subdivided into "ophthalmic origin", or "not ophthalmic origin" (i.e., cortical blindness is non-ophthalmic in origin and indicates that there is no retinal detachment or other abnormal fundus or ocular finding, except optic atrophy. Such cases will be considered central [neurologic] in origin.)
Time Frame: 18-22 Months Corrected Age
Population: Intent to Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Inositol Low Volume | Inositol Mid-level Volume | Inositol High Volume | Placebo
Number analyzed (Participants) | 24 | 24 | 23 | 27
Participants | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Gross Motor Function Greater Than or Equal to 2
Description: A Gross Motor Function Classification System (GMFCS) level of at least II (on a scale from level I to V, with I indicating normal gross motor function and higher levels indicating greater impairment). Level II is defined as Infants maintain floor sitting but may need to use their hands for support to maintain balance. Infants creep on their stomach or crawl on hands and knees with reciprocal leg movement. Infants may pull to stand and take steps holding on to furniture.)
Time Frame: 18 -22 months corrected age
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Inositol Low Volume | Inositol Mid-level Volume | Inositol High Volume | Placebo
Number analyzed (Participants) | 24 | 24 | 23 | 27
Participants | 0 | 2 | 3 | 4

ADVERSE EVENTS:
Time Frame: From start of study drug treatment through 7-days post last dose of study drug
Description: Note that the primary trial publication mislabels serious adverse events as severe adverse events.
Arm/Group | Inositol Low Volume | Inositol Mid-level Volume | Inositol High Volume | Placebo
All-Cause Mortality (participants affected / at risk) | 2/29 | 5/30 | 1/28 | 6/35
Serious Adverse Events (participants affected / at risk) | 17/29 | 20/30 | 17/28 | 28/35
Other Adverse Events (participants affected / at risk) | 24/29 | 20/30 | 19/28 | 24/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inositol Low Volume (N=29) | Inositol Mid-level Volume (N=30) | Inositol High Volume (N=28) | Placebo (N=35)
Poor perfusion or hypotension (Cardiac disorders) | 5 | 3 | 6 | 8
Delayed gastric emptying (Gastrointestinal disorders) | 3 | 7 | 5 | 7
Anemia (Blood and lymphatic system disorders) | 5 | 6 | 7 | 13
Thrombocytosis (Blood and lymphatic system disorders) | 4 | 1 | 2 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 4
Other (Renal and urinary disorders) | 0 | 0 | 0 | 2
Apnea (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 9 | 6
Other (Gastrointestinal disorders) | 3 | 0 | 2 | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inositol Low Volume (N=29) | Inositol Mid-level Volume (N=30) | Inositol High Volume (N=28) | Placebo (N=35)
Congestive heart failure (Cardiac disorders) | 0 | 1 | 0 | 0
Hypertension (Cardiac disorders) | 4 | 3 | 4 | 5
Poor perfusion or hypotension (Cardiac disorders) | 3 | 2 | 3 | 3
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Other (Cardiac disorders) | 1 | 0 | 4 | 2
Delayed gastric emptying (Gastrointestinal disorders) | 10 | 8 | 7 | 10
Direct (conjugated) hyperbilirubinemia (Gastrointestinal disorders) | 0 | 1 | 4 | 3
Elevated liver enzymes (Gastrointestinal disorders) | 3 | 1 | 0 | 1
Emesis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Other (Gastrointestinal disorders) | 2 | 1 | 0 | 2
Other (General disorders) | 1 | 0 | 1 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 7 | 4 | 4
Neutropenia (Blood and lymphatic system disorders) | 5 | 2 | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2 | 1 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 5 | 3 | 4 | 6
Other (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Infection (Infections and infestations) | 2 | 0 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 4 | 2 | 5
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2
Other (Metabolism and nutrition disorders) | 5 | 1 | 1 | 4
Apnea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 4 | 5
Increased fraction of inspired oxygen (FiO2) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Other (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0
Diuresis (Renal and urinary disorders) | 5 | 5 | 3 | 8
Elevated creatinine (Renal and urinary disorders) | 1 | 2 | 3 | 2
Elevated potassium (Renal and urinary disorders) | 1 | 2 | 1 | 1
Hematuria (Renal and urinary disorders) | 2 | 0 | 1 | 2
Oliguria (Renal and urinary disorders) | 5 | 0 | 4 | 3
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin breakdown (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators must adhere to the Neonatal Research Network Publication policies.